CLINICAL TRIAL: NCT04459117
Title: Prophylactic Treatment of the Ductus Arteriosus in Preterm Infants by Acetaminophen
Acronym: TREOCAPA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: UPCET (Unknown); PARTNERS for International clinical Research (Unknown); Connect for Children (Unknown); Global Foundation for the Care of Newborn Infants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C19-29; 2019-004297-26 (EudraCT Number)
Record Dates: First submitted 2020-06-19; First posted 2020-07-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Patency of the Ductus Arteriosus; Acetaminophen; Extreme Prematurity
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase II is a dose finding phase Phase III is a randomized, multicenter, double-blind, placebo-controlled superiority trial, two arms in a 1:1 ratio, evaluating an increasing of 10% of the percentage of survival without severe morbidity at 36 weeks of post menstrual age
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The active product is a 10 ml polyethylene ampoule of acetaminophen containing 100 mg of acetaminophen, solution for infusion, B BRAUN. The placebo product is a polyethylene ampoule of 10ml of NaCL 0.9%, B BRAUN. Polyethylene ampoule of active and placebo products are with the same appearance, in accordance with Good Manufacturing Practices Drugs for Clinical Trials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Active Comparator): The active product is a 10 ml polyethylene ampoule of acetaminophen containing 100 mg of acetaminophen, solution for infusion, B BRAUN.
  Interventions: Drug: Acetaminophen
- NaCL 0.9% (Placebo Comparator): The placebo product is a polyethylene ampoule of 10ml of NaCL 0.9%, B BRAUN. Polyethylene ampoule of active and placebo products are with the same appearance, in accordance with Good Manufacturing Practices Drugs for Clinical Trials.
  Interventions: Drug: NACL 0.9%

INTERVENTIONS:
Drug: Acetaminophen — In the 27-28 weeks gestational age group, the dosage is 2 ml/kg loading dose within 12 hours after birth followed by 0.75 ml/kg/ 6 hours during 5 days (total = 20 doses).
  In the 23-26 weeks gestational age group, the dosage will be minimum effective dose of acetaminophen to close the ductus arteriosus before or at day 7, found during the phase II.
  Arms: Acetaminophen
Drug: NACL 0.9% — In the 27-28 weeks gestational age group, the dosage is 2 ml/kg loading dose within 12 hours after birth followed by 0.75 ml/kg/ 6 hours during 5 days (total = 20 doses).
  In the 23-26 weeks gestational age group, the dosage will be minimum effective dose of acetaminophen to close the ductus arteriosus before or at day 7, found during the phase II.
  Arms: NaCL 0.9%

SUMMARY:
TREOCAPA is a Phase II/III European Multicentre study concerning the prophylactic treatment by Acetaminophen of extremely preterm infant during the first five days after birth.

The Phase II is a dose finding phase in order to assess the minimum effective dose regimen of acetaminophen for the closure of PDA for neonates with a gestational age less than 27 weeks This part of the study will be conducted in 11 NICUs, in 4 countries (France, UK, Finland and Denmark).

The Phase III is The phase III is a randomized, multicenter, double-blind, placebo-controlled superiority trial, two arms in a 1:1 ratio, evaluating an increasing of 10% of the percentage of survival without severe morbidity at 36 weeks of post menstrual age. In the intervention arm, 20 mg/kg followed by 7.5 mg/kg quarter in die (QID) will be administered to the 27-28 weeks gestational age group (dosage confirmed through PK/PD data analysis from the previous Finnian study) and the dosage selected after the conclusion of the Phase II will be administered to the 23-26 weeks gestational age group. A group sequential design, with a total of 3 analyses (2 interim analyses and a final) and the O'Brien-Fleming alpha spending function is chosen for the trial. At the same time, a Bayesian sequential analysis is planned for safety endpoints

DETAILED DESCRIPTION:
The Phase II will be conducted in 11 NICUs, in 4 countries (France, UK, Finland and Denmark). The estimated recruitment period is 6 months to enroll 30 preterm infants of 23-26 weeks of gestation. Four different loading/maintenance doses will be tested. The first level will be 20 mg/kg followed by 7.5 mg/kg quarter in die (QID) which correspond to the dosage selected for neonates with a PMA ≥27 weeks in the phase III according to data from Finland (Härkin, J Pediatr. 2016). The 2nd, 3rd and 4th level doses will stand for 25%, 50%, and 75% increase of the first level:

* 20 mg/kg loading dose then 7.5 mg/kg/6hours during 5 days (total = 20 doses)
* 25 mg/kg loading dose then 10 mg/kg/6hours during 5 days (total = 20 doses)
* 30 mg/kg loading dose then 12 mg/kg/6hours during 5 days (total = 20 doses)
* 35 mg/kg loading dose then 15 mg/kg/6hours during 5 days (total = 20 doses)

The first cohort of patients will be treated at the lowest starting dose level. Both, the Data Safety Monitoring Board (DSMB) and the statistician will be informed about the therapeutic response observed and the safety of treatment. The statistician will use these data for re-estimation of the posterior probability of success. The DSMB will be then informed about the statistical recommendation for the next dose level to use in the next cohort of 3 patients. The decision to go up, go down or stay on the same dose level will remain to the DSMB who will be free to follow or not the statistical recommendation. Dose escalation will not increase by more than one level, although dose de-escalations could be large.

At inclusion, basic data (pregnancy, blood results, birth and transfer) are recorded. After inclusion, systemic arterial pressure is measured before administration of the first dose of acetaminophen. Then the preterm infant receives a loading dose of acetaminophen. A first blood sample is collected just after end of loading dose infusion (T15min) to analyze Acetaminophen plasma level (0.2mL) ans ALT/AST (0.1ml to 0.3ml, according to local biological laboratory). Each 6 hours during the first 5 days of life, each preterm infant receives a perfusion of acetaminophen, so 20 doses are administered in total. Systemic arterial pressure is measured at 30', 60', 90', 120' after each dose. Each day, a cardiac echography is performed. After Dose 10, a second blood sample (0.3 ml to 0.5 ml according to local biological laboratory) is collected to analyze acetaminophen plasma level and ALAT & ASAT.

During visit 1 at day 3, eCRF is completed for period Day 1 to Day 3. A few "bottom of blood tubes" sampled for routine care will be kept for others acetaminophen plasma level analysis. This will be done in centres where this procedure is possible.After the last dose of acetaminophen, a blood sample of 0,3 to 0.5ml (ideally 6 hours after the start of last infusion) is collected to analyze ALAT & ASAT and Acetaminophen plasma level (0.2 ml).

During visit 2 at Day 5, eCRF is completed for period Day 4 to Day 5. A cardiac echography is performed after the last dose of acetaminophen. Data from a cerebral echography performed in routine care during the first week after the first dose will be recorded.

During Visit 3, at Day 7, CRF is completed, and the information about primary outcome (closure or not of the Ductus Arterosus) is sent by email to experts of the research unit EA 7323 " Evaluation of Therapeutics and pharmacology in perinatality and pediatrics ", University of Paris-Descartes, Paris, France.

The Phase III is a pragmatic trial. At inclusion, basic data (pregnancy, blood results, birth and transfert) are recorded. After inclusion, randomization is performed. After randomization, each infant receives a loading dose of acetaminophen or placebo before 12 hours of life. After the loading dose of Acetaminophen, a supplement of 0.1 to 0.3 ml of blood will be collected, as supplement of a blood sample performed in routine care for AST/ALT analysis. Each 6 hours during the first 5 days of life, each preterm infant receives a perfusion of placebo or acetaminophen, so 20 doses are administered in total. After the dose 10 of Acetaminophen, a supplement of 0.1 to 0.3 ml of blood will be collected as supplement of a blood sample performed in routine care for AST/ALT analysis. Few "bottom of blood tubes" sampled for routine care will be kept for acetaminophen plasma level analysis in 50 first preterm infants (25 in each gestational age group) chosen hospitalized in the NICUs participating to Phase II. This will be done in NICUs where this procedure is possible).

During visit 1 at Day 7, data describing baby care are recording day by day from Day 0 to Day 7. Around Day 7 (between Day6 and Day 10) one cardiac echography is performed.

During visit 2 at Day 28, a review of different cares received by the baby between Day 8 and Day 28 is recorded. Data from a cerebral echography performed in routine care, before 36 weeks of postmenstrual age or before discharge if it occurs before will be recorded in the eCRF. Result of the last ophthalmological examination performed in routine care before 36 weeks of postmenstrual age or before discharge if it occurs before, should be noted in the eCRF.

During visit 3 at 36 weeks of postmenstrual age or at first discharge home, whatever comes first, a review of mobidity (BPD, cerebral lesions, retinopathy, necrotizing enterocolitis) is performed to complete the primary endpoint. At the end of hospitalization, clinical data at discharge are recorded

ELIGIBILITY:
Inclusion Criteria:

* Birth between 23-26 W for Phase II, between 23-28 W for Phase III
* Post natal age < 12 hours
* Parental or Legal Authority Consent
* Parents with a social security or health insurance (if applicable according to the local regulation)

Exclusion Criteria:

* Birth defect / Congenital anomaly
* Twin-to-twin transfusion syndrome not cured
* Suspicion of pulmonary hypoplasia
* Suspicion of hepatic impairment (hemorrhagic syndrome and/or severe hypoglycemia)
* Clinical instability that can lead to rapid death
* Impossibility to start treatment before 12 hours of life
* Parents placed under judicial protection
* Participation in other clinical trial using acetaminophen during the first 5 days of life, indomethacin or ibuprofen during the first 3 days of life or using rescue treatment of PDA not recommended in the TREOCAPA trial

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 804 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Closure of Ductus Arteriosus (Primary endpoint of phase II) | Day 7
  Number of participants with closed Ductus Arteriosus (DA) assessed by echocardiography during the first 7 days of life, defined as DA closed at two consecutive echocardiographies or if the DA is closed at echocardiography of Day 7
The survival without severe morbidity (Primary endpoint of phase III) | Up to 36 weeks of post menstrual age
  the survival without severe morbidity at 36 weeks of post menstrual age or at first discharge home, whichever comes first. The severe morbidities include bronchopulmonary dysplasia (BPD Grade 3 according to NIH consensus), necrotizing enterocolitis (NEC) of Bell's stage II or III, intraventricular hemorrhage (IVH) grade III-IV or cystic leukomalacia observed at any time up to 36 weeks of post menstrual age

SECONDARY OUTCOMES:
Analgesia/sedation drugs consumption during first week after birth (Secondary endpoint of phase III) | Day 7
  Number of days during the first week the infants received sedation/analgesia treatment
Closure of Ductus arteriosus (Secondary endpoint of phase III) | Day 7
  Number of patients with a closed Ductus Arteriosus (DA) assessed by echocardiography at Day 7- Day 10
Number of back-up treatment of PDA (Secondary endpoint of phase III) | At 36 weeks of Post menstrual age
  Number of the patients receiving back-up treatment
Number of days during the first week after birth with catecholamines administration (Secondary endpoint of phase III) | Day 7
  Number of days during the first week the infants received catecholamines in perfusion
Early pulmonary hemorrhage (Secondary endpoint of phase III) | Day 7
  Number of infants with early pulmonary hemorrhage
Blood acetaminophen levels in extrem preterm infant (Secondary endpoint of Phase II and Phase III) | Day 7
  Analysis of acetaminophen levels according to the administered dose and the time of sample collection
Toxicity of Acetaminophen in extrem preterm infant (Secondary endpoint of Phase II and Phase III) | Day 7
  Number of patient with increase of AST/ALT more than 2 times the normal value (according to local standards) or the first AST/ALT dosage before loading dose of Acetaminophen if if available in standard care

CONTACTS AND LOCATIONS:
Locations (36):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium
- The Juliane Marie Centre, Rigshospitalet, Copenhagen University hospital, Copenhagen, Denmark
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - Tallinn Children's Hospital, Tallinn
  - Tartu University Hospital, Neonatal and Paediatric Intensive Care Unit, Tartu
- Finland (5):
  - Helsinki University Hospital, Department of Children and Adolecents, Neonatology, Helsinki
  - Kuopio University Hospital, Department of Pediatrics, Kuopio
  - Oulu University Hospital, Department of Pediatrics, Oulu
  - Tampere University Hospital, Department of Pediatrics, Tampere
  - Turku University Hospital, Department of Peadiatrics, Turku
- France (16):
  - CHU Angers, Angers
  - Hopital Jeanne de Flandre, Lille
  - Hôpital Croix-Rousse, Lyon
  - Hospice civils de Lyon, Hopital Femme Enfant, Lyon
  - Hôpital Marseille Nord, Marseille
  - Hôpital de la conception, Marseille
  - Hôpital Arnaud de Villeneuve, Département de Pédiatrie Néonatale et Réanimation Pédiatrique, Montpellier
  - CHU Nantes, Hopital mére Enfant, Nantes
  - Hôpital Necker - Enfants malades, Paris
  - CENTRE hospitalier intercommunal de Creteil, Paris
  - Hopital Cochin, Service de Médecine et Réanimation néonatales de Port-Royal, Paris
  - Hopital Robert Debré, Néonatologie, Paris
  - CHU Rennes, Hopital Sud, Rennes
  - CHU Strasbourg, Hôpital de Hautepierre, Strasbourg
  - Centre Hospitalo-Universitaire de Toulouse, Toulouse
  - CHRU de Tours, Tours
- Bács Kiskun COUNTY HOSPITAL, Kecskemét, Hungary
- Cork University Hospital, Cork, Ireland
- Azienda Ospedaliero - Universitaria delle Marche, Ancona, Italy
- Oslo University Hospital, Oslo, Norway
- Portugal (2):
  - Centro Hospitalar Universitário Lisboa Norte, EPE -Hospital Santa Maria, Lisbon
  - Centro Hospitalar e Universitário do Porto, EPE - Centro Materno Infantil do Norte, Porto
- Karolinska University Hospital, Solna, Sweden
- Switzerland (3):
  - Hopital Universitaire de Geneve (HUG) - Hopital des enfants, Geneva
  - University Children's Hospital Lausanne, Lausanne
  - University Hospital of Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ursino M, Alberti C, Cambonie G, Kemp R, Vanhecke A, Levoyer L, Diallo A, Hallman M, Roze JC; TREOCAPA study group. TREOCAPA: prophylactic treatment of the ductus arteriosus in preterm infants by acetaminophen-statistical analysis plan for the randomized phase III group sequential trial. Trials. 2025 Feb 13;26(1):52. doi: 10.1186/s13063-025-08751-8. PMID 39948605
- [Derived] Bouazza N, Cambonie G, Flamant C, Rideau A, Tauzin M, Patkai J, Gascoin G, Lumia M, Aikio O, Lui G, Bournaud LF, Walsh-Papageorgiou A, Tortigue M, Baruteau AE, Kallio J, Hallman M, Diallo A, Levoyer L, Treluyer JM, Roze JC. Prophylactic Intravenous Acetaminophen in Extremely Premature Infants: Minimum Effective Dose Research by Bayesian Approach. Paediatr Drugs. 2024 Jan;26(1):83-93. doi: 10.1007/s40272-023-00602-w. Epub 2023 Nov 17. PMID 37978159